CLINICAL TRIAL: NCT04009265
Title: Multicenter Prospective Randomized Controlled Study of Adjuvant Chemotherapy, Chemoradiotherapy and Surgery Alone in the Treatment of pN1-2 (pT1b-3N1-2M0) Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Study Compare Adjuvant Chemotherapy, Chemoradiotherapy and Surgery Alone for pN1-2(pT1b-3N1-2M0) Esophageal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACRTEC UNION
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; adjuvant chemotherapy; adjuvant chemoradiotherapy; surgery
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chemotherapy (Experimental): Docetaxel 75mg/m2, 3w, 2cycles. DDP 75mg/m2, 3wl, 2cycles.
  Interventions: Combination Product: adjuvant treatment
- Chemoradiotherapy (Experimental): 5040cGy, 180cGy/d, 28F Concurrent Docetaxel 60mg/m2, 3w, 2cycles DDP 60mg/m2, 3w, 2cycles
  Interventions: Combination Product: adjuvant treatment
- Surgery alone (No Intervention): Surgery alone, no adjuvant treatment.

INTERVENTIONS:
Combination Product: adjuvant treatment — adjuvant treatments include chemotherapy or chemoradiotherapy
  Arms: Chemoradiotherapy; Chemotherapy

SUMMARY:
A multi-center prospective randomized controlled study was conducted to compare the effects of adjuvant chemotherapy, chemoradiotherapy and surgery alone for the patients with esophageal cancer.

DETAILED DESCRIPTION:
A multi-center prospective randomized controlled study was conducted to compare the effects of adjuvant chemotherapy, chemoradiotherapy and surgery alone on the overall survival rate (OS) and disease-free survival (DFS) of patients with pN1-2 (pT1b-3N1-2M0) thoracic esophageal squamous cell carcinoma, and to observe the safety, side effects of adjuvant therapy and the impact on the quality of life of patients after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants volunteer to participate the study and signed the informed consent.
2. Surgical methods: Radical resection of tumors (R0) was performed, and pathological examination confirmed the diagnosis of thoracic esophageal squamous cell carcinoma.
3. No antineoplastic treatments before operation.
4. According to the 8th edition of AJCC staging, pN1-2 (pT1b-3N1-2M0) stage of esophageal cancer;
5. WHO PS score: 0-1;
6. Age and gender: 18-75 years old, male and female unlimited;
7. Laboratory examination within one week before the adjuvant treatment confirmed that the cardiac, hepatic and renal functions met the requirements.

Exclusion Criteria:

1. The surgical approach is left thoracic approach;
2. Patients with severe postoperative complications who cannot receive adjuvant therapy;
3. Received other anti-tumor treatment before enrollment; At the same time, patients with malignant tumors of other sites were excluded, except non-melanoma skin cancer, in-situ cervical cancer or cured early prostate cancer.
4. Abnormal coagulation function, bleeding tendency (such as active gastrointestinal ulcer) or receiving thrombolytic or anticoagulant treatment;
5. Patients with original severe heart disease, including congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction within half a year, severe heart valve disease and intractable hypertension; Severe hepatic and renal insufficiency;
6. Patients with uncontrollable neurological, mental illness or mental disorder, poor compliance, and inability to cooperate or describe treatment response;
7. Known or suspected allergy to chemotherapeutic drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3-year overall survival
  overall survival rate of each arms
Overall Survival | 5-year overall survival
  overall survival rate of each arms

SECONDARY OUTCOMES:
Disease Free Survival | 3-year disease free survival
  Disease free survival rate of each arms
Disease Free Survival | 5-year disease free survival
  Disease free survival rate of each arms
Adverse Events | 1 year
  Number and degree of Adverse Events based on Common Toxicity Criteria for Adverse Effects(CTCAE)
Scores of Quality of Life | 5 years
  Assess the quality of life based on EORTC QLQ-C30 and OES18

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, MD, Study Director — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No